CLINICAL TRIAL: NCT03766633
Title: Accuracy of Established Manual Versus New Semi-automated Liver Volumetry Software in Patients Undergoing Living Donor Liver Transplantation
Brief Title: Accuracy of the LiverVision® Semi-automated Liver Volumetry Software
Acronym: LiverVision
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Ankara University (Other); University Hospital Tuebingen (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Dimitri Raptis, Principal Investigator, Royal Free Hospital NHS Foundation Trust
Other Study IDs: LV.2018.04.29
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Liver Diseases; Liver Cancer
Keywords: LiverVision; Liver; Volumetry; Semi-automated; Living donor liver transplantation; Surgery
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Living liver donors: This is a group of living liver donors that underwent a CT prior to donating their partial liver to a recipient.
  Interventions: Diagnostic Test: Liver volumetry of the graft on CT

INTERVENTIONS:
Diagnostic Test: Liver volumetry of the graft on CT — Preoperative liver volumetry using the CT images of the potential living liver donors.

SUMMARY:
The LiverVision® software was designed to provide three-dimensional (3D) visualisation of the liver using Computed Tomography (CT) scans. It provides semi-automated volumetry measurements, vascular structure and territory tools.

DETAILED DESCRIPTION:
Liver volumetry has been widely used in liver surgery and living donor liver transplantation to estimate the future liver remnant or the required liver volume for the recipient, respectively.

Liver volumetry is typically performed using CT imaging with specially designed software. Such manual measurements are time consuming and there is an ongoing debate whether the they reflect the actual liver volume when performed by radiologists or surgeons as well as according to the different software currently available in the market.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Living liver donors.

Exclusion Criteria:

* Recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive living liver donors that underwent a CT prior to liver donation. The raters will be 6 surgeons and 6 radiologists, both junior and senior.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2018-04-29 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the LiverVision® software volumetric measurements | Baseline (CT performed prior to donation).
  Accuracy of the LiverVision® software volumetric measurements assessed by correlation and agreement statistics with the manual volumetric measurements as well as the actual graph weight (reference standard).

SECONDARY OUTCOMES:
Learning curve of the raters | Baseline (CT performed prior to donation).
  Assessment of the learning curve of the raters when using LiverVision® software assessed by the time required for the volumetric measurements and the accuracy of the results.
Certainty and accuracy of the volumetric measurements. | Baseline (CT performed prior to donation).
  Correlation of the degree of certainty of the raters with the accuracy of their volumetric measurements.
Comparison | Baseline (CT performed prior to donation).
  Comparison of the accuracy among junior, senior, surgeons and radiologists (4 groups)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Malago', MD, PhD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (3):
- Universitätsklinikum Tübingen, Tübingen, Germany
- Ankara Üniversitesi Tıp Fakültesi Cebeci Araştırma ve Uygulama Hastanesi, Ankara, Turkey (Türkiye)
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing individual participant data.

REFERENCES:
- See also: Data management platform for the LiverVision.org Study — https://LiverVision.org/
- See also: Cloud Graphical User Interface for R Statistics, the statistical analysis software — https://rBiostatistics.com/